CLINICAL TRIAL: NCT01948817
Title: A Prospective Single Arm Study to Assess the Efficacy and Safety of Deferasirox 20 mg/kg BID in Transfusion Dependent Thalassemia Patients Inadequately Responding to Current Treatment With Doses > 35mg/kg QD (Once a Day).
Brief Title: Deferasirox BID (Twice a Day) in Transfusion Dependent Thalassemia Patients With Inadequate Response to High Doses
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670A2420; 2013-002624-16 (EudraCT Number)
Record Dates: First submitted 2013-09-19; First posted 2013-09-24 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2014-01

CONDITIONS: Focus on Transfusion Dependent Thalassemia Patients Who Are Inadequate Responders to Deferasirox > 35mg/kgQD
Keywords: Thalassemia
MeSH Terms: conditions — Thalassemia | interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Deferasirox (Experimental): Deferasirox 20mg/kg taken BID
  Interventions: Drug: Deferasirox

INTERVENTIONS:
Drug: Deferasirox — Deferasirox 20mg/kg taken BID

SUMMARY:
This is an open label, single arm, and multicenter study. The study will include the following phases. A screening phase which lasts for 4 weeks to determine patient eligibility. This phase will be followed by a 24 week Open label treatment phase. The study treatment is defined as deferasirox 20mg/kg BID 9Twice a day). Serum Ferritin Levels and MRI (Magmetic Resonance Imaging) LIC (Liver Iron Concentration) will be measured to evaluate the response to BID.

DETAILED DESCRIPTION:
Study treatment is defined as deferasirox 20 mg/kg BID. The study treatment duration is 24 weeks. After the baseline visit, patient visits will occur weekly during the first month because key safety parameters need to be performed weekly in the first month of treatment and then every 4 weeks thereafter until week 24 End of Treatment (EOT).

Patients will have their first dose of study treatment at Visit 3. Safety assessments are routinely performed including collection of AEs (Adverse Events), SAEs (Serious ADverse Events<, vital signs, physical examination, ECG (Electrocardiograph), hematological and biochemistry assessments.

Patients will continue therapy until intolerable toxicity, patient decision or after 24 weeks treatment duration at which point and End of Treatment (EOT) visit will be performed and the End of Treatment CRF( Case Report Form) will be completed.

30 day Safety follow-up Patients who discontinue study drug before completing the study should be scheduled for a visit as soon as possible, at which time all of the assessments listed for the final visit will be performed. At a minimum, all patients who discontinue study treatment, including those who refuse to return for a final visit, will be contacted for safety evaluations during the 30 days following the last dose of study drug.

All patients must be followed for AEs and SAEs that may have occurred after discontinuation from the study treatment. The safety follow-up visit will take place 30 days after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained prior to any screening procedures
* Male or female aged ≥ 2 years at screening
* Patients with transfusion dependent thalassemia
* Patients confirmed as inadequate- responders to deferasirox > 35 mg/kg QD and treated with QD for at least 6 months
* Regular transfusion indicated by a blood requirement ≥ 8 blood transfusions per year at screening
* Serum ferritin level > 2,500 ng/mL at screening (two consecutive values at least 2 weeks apart from each other)
* One SF measurement > 2,500 ng/mL between 6 and 9 months prior to study enrollment
* Three SF measurements > 2,500 ng/mL, performed at least 3 weeks apart from each other, during the 6 month treatment with QD dosing of deferasirox prior to study enrollment
* The average of the two screening SF values (collected 2 weeks apart from each other) must not show a decrease from the 6 to 9 month SF value taken prior to study enrollment
* The average of the two screening SF values (collected 2 weeks apart from each other) must not show a decrease from each of the three SF values obtained during the 6 months of deferasirox QD treatment prior to study enrollment
* LIC ≥ 7 mg Fe/g dw measured at the screening visit, (this value will be used as a baseline measurement

Exclusion Criteria:

* Patients who are intolerant to > 35 mg/kg/day QD of deferasirox in the 6 months prior to study enrollment
* Patients with mean levels of ALT >5 x ULN
* Patients with serum creatinine above the upper limit of normal (ULN)
* Significant proteinuria as indicated by a urinary protein/creatinine ratio > 0.5 (mg/mg)
* Creatinine clearance ≤ 60 ml/min
* Chronic hepatitis B infection, active hepatitis C infection
* History of a positive HIV test
* Uncontrolled systemic hypertension
* Patients participating in another clinical trial or receiving a systemic investigational drug within the past 4 weeks or topical investigational drug within the past 7 days of screening
* History of non-compliance with medical regimens or patients who are considered potentially unreliable and/or not cooperative, unwilling or unable to comply with the protocol
* History of hypersensitivity to any of the study drug or excipients
* Significant medical condition interfering with the ability to partake in this study (e.g. systemic uncontrolled hypertension, unstable cardiac disease not controlled by standard medical therapy, systemic disease (cardiovascular, renal, hepatic etc.)
* History of drug or alcohol abuse within the 12 months prior to enrollment.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Mean relative change in SF (Serum Ferritin) | Baseline, 24 Weeks
  To evaluate the efficacy of a twice-daily dose regimen of deferasirox in inadequate-responders to a once daily dose regimen as measured by relative change in serum ferritin from baseline to 24 weeks of treatment

SECONDARY OUTCOMES:
Mean Absolute/relative change in LIC | Baseline, 24 Weeks
  To evaluate the efficacy of BID deferasirox in liver iron removal as measured by MRI by absolute/relative change from baseline to 24 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals